CLINICAL TRIAL: NCT07161128
Title: Pedobarographic Evaluation of Gait Biomechanics in Patients Treated With Arthroscopic Microfracture and Biologic Cartilage Scaffold for Osteochondral Defect (OCD) of Talus
Brief Title: Gait Pattern Analysis After Arthroscopic Treament of Osteochondral Defects of Talus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Furkan ARAL, Chief Resident in Orthopaedic Surgery, Principal Investigator, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gazi University Hospital
Record Dates: First submitted 2025-06-16; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Osteochondral Defects of Talus; Gait Analysis; Microfracture Procedure; Biological Scaffold
Keywords: pedobarography; gait analysis; ocd of talus; microfracture
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microfracture + Biologic Scaffold (Experimental)
  Interventions: Procedure: arthroscopic microfracture and biological scaffold implementation for osteochondral defects of talus

INTERVENTIONS:
Procedure: arthroscopic microfracture and biological scaffold implementation for osteochondral defects of talus — All enrolled patients will undergo a standardized single-stage arthroscopic procedure under spinal or general anesthesia with the patient supine and the ankle placed in appropriated position. Standard anteromedial and anterolateral portals are established. The talar osteochondral defect is inspected, measured, and any unstable cartilage is sharply débrided to create stable vertical walls, exposing healthy subchondral bone. Using a 1.0- to 1.2-mm awl, multiple perforations are made perpendicular to the lesion base, 3-4 mm apart and ~2-4 mm deep, until uniform "marrow fat-bleeding" is observed-mobilizing mesenchymal stem cells .A sterile, resorbable, type-I/III collagen bilayer scaffold is trimmed to the exact defect footprint using a template fashioned intra-operatively.

SUMMARY:
The study will investigate alterations in post-surgical gait patterns among patients who have undergone all arthroscopic microfracture and biological scaffold implementation surgery for the osteochondral lesions of talus. The gait biomechanics of patients scheduled for surgery will be assessed preoperatively using pedobarographic analysis. Subsequent changes in walking biomechanics will be evaluated and interpreted at the 6th postoperative months. Consequently, the impact of the all arthroscopic treatment of osteochondral lesions of talus on walking will be documented.

DETAILED DESCRIPTION:
Osteochondral defects (OCDs) of the talus are lesions that extend into the subchondral bone. They most commonly occur after ankle fractures, dislocations, or other ankle injuries. Spontaneous necrosis, systemic vascular disorders, and metabolic diseases have also been implicated in the development of talar OCD.

Current treatment strategies-selected according to lesion size, location, and patient characteristics-range from conservative modalities (weight-bearing restriction, NSAIDs, immobilization) to arthroscopic debridement, bone marrow-stimulating techniques such as microfracture or nanofracture combined with biologic scaffolds, autologous chondrocyte-based procedures (ACI, MACI, AMIC), autologous osteochondral transfers (mosaicplasty/OAT), and more recently, biologic augmentations with platelet-rich plasma (PRP) or bone marrow aspirate concentrate (BMAC).

The microfracture technique is usually performed arthroscopically. Perforation of the subchondral plate recruits mesenchymal stem cells that drive cartilage repair. Concomitant use of a biologic scaffold has been shown to enhance cartilage regeneration and improve functional scores. While microfracture provides an initial stimulus for defect filling, biologic cartilage scaffolds support cell adhesion and foster the formation of hyaline-like tissue. Autologous osteochondral transfers are preferred for larger lesions, and among autologous chondrocyte-based techniques, no meaningful short-term clinical differences have been demonstrated.

Plantar pressure analysis (pedobarography) yields objective information on foot and ankle biomechanics during gait and is widely used to detect changes after orthopedic surgery. By quantifying plantar pressure distribution, pedobarography enables detailed assessment of foot and ankle loading patterns. In patients with talar OCD, gait analyses have shown that the ankle tends to assume a valgus position during walking; medial talar lesions are associated with reduced plantarflexion at the Lisfranc joint, whereas lateral talar lesions demonstrate increased midfoot peak pressure.

This study will evaluate postoperative changes in gait biomechanics-measured by pedobarography-in patients with talar OCD treated arthroscopically with microfracture and a biologic cartilage scaffold. We hypothesize that the abnormal plantar pressure distribution observed preoperatively will normalize after surgery, bringing gait biomechanics closer to those of healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* presence of osteochondral defect on talus confirmed with MRI
* planning for arthroscopic microfracture+ biological scaffold surgery

Exclusion Criteria:

* presence of foot and ankle deformities
* Presence of orthopedic or neurological pathologies that may affect walking biomechanics.
* History of prior foot and ankle surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Peak Plantar Pressure (kPa) in Pedobarographic analysis | Baseline (1 day before surgery) and 6 months after surgery
  Peak plantar pressure will be assessed using a computerized pedobarographic platform equipped with pressure sensors and dedicated gait analysis software. Patients will walk barefoot at a self-selected, comfortable speed with arms relaxed at the sides, following a natural gait. In each session, five valid gait trials will be recorded. For each trial, the maximum plantar pressure value under the entire foot during stance will be extracted. The mean value of the five trials will be reported. This outcome quantifies the highest load experienced by the plantar surface during walking and will allow comparison of preoperative and postoperative gait biomechanics.
Plantar Pressure-Time Integral (kPa·s) in Pedobarograpic Analysis | Baseline (1 day before surgery) and 6 months after surgery
  The plantar pressure-time integral will be measured using the same pedobarographic platform. During dynamic gait analysis, patients will complete five valid walking trials at a natural speed. For each trial, the cumulative pressure applied over time to the plantar surface during the stance phase will be calculated and expressed as kPa·s. The average of the five trials will be reported. This measure reflects the duration and magnitude of plantar loading and provides information on changes in gait mechanics following surgery.
Plantar Contact Area (cm²) in Pedobarographic Analysis | Baseline (1 day before surgery) and 6 months after surgery
  Plantar contact area will be evaluated using the pedobarographic platform during dynamic gait analysis. Patients will walk at a self-selected speed, and five valid gait trials will be collected. For each trial, the total plantar surface area in contact with the platform during stance will be computed and expressed in square centimeters. The mean of the five trials will be reported. This outcome reflects how much of the plantar surface participates in load transfer during walking and will be used to assess functional improvement after surgery.
Center of Pressure Excursion Index (%) in Pedobarographic Analysis | Baseline (1 day before surgery) and 6 months after surgery
  The Center of Pressure (COP) Excursion Index will be calculated from dynamic pedobarographic recordings. Patients will walk barefoot at a self-selected, comfortable speed, with five valid gait trials collected per session. The COP trajectory during stance will be analyzed, and the mediolateral deviation of the COP path will be expressed as a percentage relative to foot width (Excursion Index). The average value from the five trials will be reported. This outcome reflects dynamic postural control and foot loading patterns during gait and will be compared between the preoperative and postoperative assessments.Baseline (1 day before surgery) and 6 months after surgery

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS) | Baseline (1 day before surgery) and 6 months after surgery
  The hindfoot score comprises nine questions that assess pain, function, and alignment. Within the survey, one question pertains to pain, seven questions address function, and one question relates to alignment. The pain section is appraised on a scale of 40 points, the function section on 50 points, and the alignment section on 10 points, summing up to a total of 100 points. A higher score indicates better functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Petersen T, Gordon JA, Kant A, Fava M, Rosenbaum JF, Nierenberg AA. Treatment resistant depression and axis I co-morbidity. Psychol Med. 2001 Oct;31(7):1223-9. doi: 10.1017/s0033291701004305. PMID 11681548
- [Background] Giannini S, Buda R, Cavallo M, Ruffilli A, Cenacchi A, Cavallo C, Vannini F. Cartilage repair evolution in post-traumatic osteochondral lesions of the talus: from open field autologous chondrocyte to bone-marrow-derived cells transplantation. Injury. 2010 Nov;41(11):1196-203. doi: 10.1016/j.injury.2010.09.028. Epub 2010 Oct 8. PMID 20934692
- [Background] Ramponi L, Yasui Y, Murawski CD, Ferkel RD, DiGiovanni CW, Kerkhoffs GMMJ, Calder JDF, Takao M, Vannini F, Choi WJ, Lee JW, Stone J, Kennedy JG. Lesion Size Is a Predictor of Clinical Outcomes After Bone Marrow Stimulation for Osteochondral Lesions of the Talus: A Systematic Review. Am J Sports Med. 2017 Jun;45(7):1698-1705. doi: 10.1177/0363546516668292. Epub 2016 Nov 16. PMID 27852595
- [Background] Steadman JR, Briggs KK, Rodrigo JJ, Kocher MS, Gill TJ, Rodkey WG. Outcomes of microfracture for traumatic chondral defects of the knee: average 11-year follow-up. Arthroscopy. 2003 May-Jun;19(5):477-84. doi: 10.1053/jars.2003.50112. PMID 12724676
- [Background] Migliorini F, Eschweiler J, Maffulli N, Schenker H, Driessen A, Rath B, Tingart M. Autologous Matrix Induced Chondrogenesis (AMIC) Compared to Microfractures for Chondral Defects of the Talar Shoulder: A Five-Year Follow-Up Prospective Cohort Study. Life (Basel). 2021 Mar 16;11(3):244. doi: 10.3390/life11030244. PMID 33809441
- [Background] Cheng L, Wang X. Advancements in the treatment of osteochondral lesions of the talus. J Orthop Surg Res. 2024 Dec 6;19(1):827. doi: 10.1186/s13018-024-05314-6. PMID 39639331
- [Background] Gianakos AL, Yasui Y, Hannon CP, Kennedy JG. Current management of talar osteochondral lesions. World J Orthop. 2017 Jan 18;8(1):12-20. doi: 10.5312/wjo.v8.i1.12. eCollection 2017 Jan 18. PMID 28144574
- [Background] Ferkel RD, Zanotti RM, Komenda GA, Sgaglione NA, Cheng MS, Applegate GR, Dopirak RM. Arthroscopic treatment of chronic osteochondral lesions of the talus: long-term results. Am J Sports Med. 2008 Sep;36(9):1750-62. doi: 10.1177/0363546508316773. PMID 18753679